CLINICAL TRIAL: NCT05765019
Title: Investigation of the Efficiency of Spinal Mobilization in Patients With Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Eylem KÜÇÜK, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HacettepeUE
Record Dates: First submitted 2023-02-19; First posted 2023-03-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; Core stabilization exercises; Spinal mobilization; Manual therapy; Pulmonary function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal mobilization group (Experimental)
  Interventions: Other: Spinal mobilization; Other: Core stabilization exercise
- Core stabilization exercise group (Active Comparator)
  Interventions: Other: Core stabilization exercise

INTERVENTIONS:
Other: Spinal mobilization — Spinal mobilization and core stabilization exercise
  Arms: Spinal mobilization group
Other: Core stabilization exercise — Stabilization exercises for the spine

SUMMARY:
In this study, it was aimed to evaluate the effect of spinal mobilization techniques applied in addition to core stabilization exercises in Adolescent Idiopathic Scoliosis (AIS) patients.

Consecutive adolescents with idiopathic scoliosis, aged 10 to 16 years, without a brace, and with a Cobb curvature of 10 to 25 degrees were randomly divided into two groups using the closed envelope method: Spinal mobilization and core stabilization exercise were applied to the experimental group; Only core stabilization exercises were applied to the control group.

Both groups received interventions twice a week for 10 weeks. Outcome measurements were made before treatment and after 10 weeks of treatment.

DETAILED DESCRIPTION:
This study was a randomized controlled trial in which participants and assessor were blinded. This study was carried out in Amasya University Ruhi Tingiz Physical Therapy and Rehabilitation Hospital Rehabilitation Unit between August 2022 and January 2023. Ethics committee approval was obtained from Amasya University (E-76988455-050.01.04-83314) on 05.08.2022 to conduct the study. Before the study, face-to-face interviews were conducted with the all participants and parents and informed about the subject and purpose of the study. Verbal and written consent was obtained from the all participants and parents.

Sample size: The sample of the study was calculated with the G*Power 3.1 program, and the effect size (d=1.0) was calculated according to the double-tailed hypothesis method, taking into account the study. (d=1.0; α=0.05; 1-ß=0.80). Confidence interval was determined as 80% and margin of error was 5% (α=0.05). As a result of the calculation, it was determined that there should be 17 adolescent scoliosis patients for the control group, 17 for the experimental group, and a total of 34 adolescent scoliosis patients. Considering the possible data losses of the participants, we planned to include a total of 40 participants, 20 in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIS
* Age 10-16 years
* Cobb angle was between 10° and 25
* Risser sing did not exceed 4
* Informed consent forms were signed by the parents and children

Exclusion Criteria:

* Used brace,
* Had previous spinal surgery, inferior limb length difference,
* Could not exercise due to another injury/diagnosis,
* Had neuromuscular, psychiatric, cardiovascular, respiratory insufficiency and mental disability

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Cobb angle | Change from pretreatment and 10 weeks after treatment.
  The most accepted way of scoliosis evaluation is Cobb angle measurement performed on frontal plane x-ray. The Cobb angle is the curvature of the spine, and measuring it is essential for determining the severity of scoliosis, selecting the best course of action, and monitoring the progression or regression of cases following treatment. The Cobb angle measure as the vertically intersecting angle after determining the vertebrae above the apex and below the apex, which are the most tilted from the concave side of the curvature of the spine.

SECONDARY OUTCOMES:
Angle of Trunk Rotation | Change from pretreatment and 10 weeks after treatment.
  It assessed with a Bunnell scoliometer is a type of inclinometer that measures the asymmetry of the degree of axial rotation on both sides of the body. Assessment is in a standing, forward-bending position bent-over position (arms dangling, palms pressed together) with the pelvis horizontal, and subject standing on a foot template
Pulmonary Functions Test- PEF (Peak expiratory flow) | Change from pretreatment and 10 weeks after treatment.
  Peak expiratory flow (PEF) is the volume of air forcefully expelled from the lungs in one quick exhalation, and is a reliable indicator of ventilation adequacy as well as airflow obstruction.
Pulmonary Functions Test- FEV1 (Forced expiratory volume in the first second) | Change from pretreatment and 10 weeks after treatment.
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration
Pulmonary Functions Test-FVC (Forced vital capacity) | Change from pretreatment and 10 weeks after treatment.
  Forced vital capacity, the maximum amount of air you can forcibly exhale from your lungs after fully inhaling.
Pulmonary Functions Test- FEV1/FVC | Change from pretreatment and 10 weeks after treatment.
  The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs.
Walter Reed Visual Assessment Scale | Change from pretreatment and 10 weeks after treatment.
  It was designed to measure physical deformity as perceived by patients with idiopathic scoliosis. The scale assesses seven aspects of the deformity: spinal curvature, rib prominence, flank prominence, deformity/alignment of the thorax with respect to the pelvis, trunk imbalance, shoulder asymmetry and scapular asymmetry. Scores for each catagory range from 1 (no deformity) to 5 (the worst deformity), and the total score is generated from the sum of the scores from the seven domains.
Scoliosis Research Society-22 | Change from pretreatment and 10 weeks after treatment.
  Scale is a simple and practical quality of life questionnaire specially created for individuals with scoliosis. SRS includes parameters such as pain, self-image/appearance, function/activity, mental health, and satisfaction with treatment. It is also stated that it is effective in evaluating the changes that occur with treatment. The questionnaire has a total of 22 items that are scored from 1 (worst) to 5 (best) for each item.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)